CLINICAL TRIAL: NCT06133855
Title: Impact of Electromagnetic Field Therapy on Pain Severity and Functional Disability in Patients With Mechanical Back Pain: a Randomized Controlled Trial
Brief Title: Impact of Electromagnetic Field Therapy on Pain and Function in Patients With Mechanical Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HAPO-06-B-001; ECM#2023-2104
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Mechanical Low Back Pain
Keywords: Electromagnetic Field; Mechanical back pain; Myofascial trigger point; Pain severity
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Intervention Model Description: pulsed electromagnetic fields therapy and traditional physical therapy program
Who Masked: Investigator, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed electromagnetic field (Experimental): the patients will receive pulsed electromagnetic field plus traditional physical therapy program three times a week for four weeks
  Interventions: Radiation: Pulsed electromagnetic field; Other: traditional physical therapy program
- traditional physical therapy program (Active Comparator): the patients will receive traditional physical therapy program three times a week for four week
  Interventions: Other: traditional physical therapy program

INTERVENTIONS:
Radiation: Pulsed electromagnetic field — The experimental group will be treated with an ASA magnetic field device (Automatic PMT Quattro Pro) at a frequency of 50 Hz in addition to the traditional physical therapy program. Each session will consist of 20 minutes of the patient lying prone and exposed to low-intensity 20-gauss PEMF.
  Arms: Pulsed electromagnetic field
Other: traditional physical therapy program — A traditional physical therapy program will include
  Infrared radiation for 20 minutes per session for 3 sessions per week for 4 weeks
  Ultrasonic: 1 MHz; continuous mode of application: 1.5 w/cm2 for 5 minutes; 3 sessions per week for 4 weeks.
  stretching exercises for the hamstring, calf muscles, and back muscles. 3 sessions per week for 4 weeks
  Strengthening exercises for back and abdominal muscles.

SUMMARY:
This study aims to investigate the impact of electromagnetic field therapy on pain severity and functional disability in mechanical back pain patients suffering from myofascial trigger points.

DETAILED DESCRIPTION:
Lower back pain, or LBP, is a major global health issue that affects functioning, social participation, and personal financial prosperity on a variety of biophysical, psychological, and social levels. In today's industrial society, it impacts roughly 50-80% of people who are of working age. Mechanical back pain patients suffer from myofascial trigger points (MTrPs), which are classified as either active or latent. Activated MTrPs cause either sudden onset of pain or in response to movement, stretching, or compression. Latent MTrPs are typically symptom-free, but when squeezed, they can re-create pain or irritation. Muscle weakness and limited ROM are other common signs of mechanical back pain, along with local as well as referred pain that affect patients functional activities.

Recently, there has been a focus on non-pharmacotherapy for low back pain. One of them is electromagnetic field therapy (PEMF) which uses electromagnetic field pulses to stimulate tissue healing without causing heat damage to the tissue. The FDA has given electromagnetic field therapy devices approval for treating post-operative pain, swelling, and osteoarthritis. Furthermore, PEMF devices are frequently used to treat bone fractures, inflammation, arthritis, pain, swelling, and chronic wounds.

Thus, the purpose of this study is to ascertain how electromagnetic field therapy affects the degree of pain and functional impairment in mechanical back pain patients suffering from myofascial trigger points.

ELIGIBILITY:
Inclusion Criteria:

1. The patients age from 20 to 40 years for both genders.
2. Patients (office worker) with mechanical back pain for 3 months ago and has not been diagnose as a specific disease or spinal abnormality.
3. Patients suffering from active MTrPS in lower back muscles.
4. The study patients must be willing to participate in the study.

Exclusion Criteria:

1. Neurological, systemic illness and infectious diseases such as rheumatologic diseases, tumor.
2. Psychiatric/mental deficit.
3. Patients who had a previous surgical history (within 6 months) were also excluded prior to the baseline assessment.
4. Vertebral compression fracture
5. Pregnancy and lactation.
6. Existing lower limb symptoms.
7. Cardiopulmonary disorders with reduced activity tolerance. -

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  A Visual Analogue Scale (VAS) will be used by the patient to mark his or her level of pain, usually 10 cm long, ranging from no pain or discomfort (zero) to the worst pain that the patient can possibly feel.

SECONDARY OUTCOMES:
functional disability | up to four weeks
  Arabic version of Oswestry Disability Index will be used for assessment of functional disability
lumbar flexion and extension assessment | up to four weeks
  modified-modified Schober test will be used to assess lumbar flexion and extension
lumbar lateral flexion assessment | up to four weeks
  tape measurement will be used to assess lumbar lateral flexion

CONTACTS AND LOCATIONS:
Overall Officials: Ghada MR Koura, Ass. prof, Study Director — King Khalid University, Saudi Arabia
Locations (1):
- Ghada Mohamed Rashad Koura, Abhā, Saudi Arabia